CLINICAL TRIAL: NCT02285985
Title: Effects of Saxagliptin on Adipose Tissue Inflammation in Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 032; 0086 (Other: Phoenix VA Health Care System)
Record Dates: First submitted 2014-06-17; First posted 2014-11-07 (Estimated); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Adipose tissue; Inflammation; .Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Obesity | interventions — saxagliptin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin (Experimental): Saxagliptin (trade-name ONGLYZA™) is used along with diet and exercise to lower blood sugar levels in patients with Type II diabetes (condition in which blood sugar is too high because the body does not produce or use insulin normally). Saxagliptin is in a class of medications called dipeptidyl peptidase-4 (DPP-4) inhibitors. It works by increasing the amount of insulin produced by the body after meals when blood sugar is high As the blood sugar returns towards normal, the medication effect on insulin is decreased.
  Interventions: Drug: Saxagliptin
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — Tablets: 5 mg
  Other Names: ONGLYZA™; Inhibitor
  Arms: Saxagliptin
Drug: Placebo — Tablets: 5mg
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
In this research study, Investigators will be comparing the effects of a medication Saxagliptin versus placebo (a similar looking pill that contains no medication) on inflammation in the body.

Research Hypothesis DPP-4 inhibition by saxagliptin (ONGLYZA™) reduces adipose tissue inflammation in obese individuals and this is characterized by decreases in a) reactive oxygen species (ROS) production, b) toll-like receptors (TLR) and NF-kappa B pathway activation, c) expression of pro-inflammatory genes, d) macrophage infiltration, and e) secretion of pro-inflammatory factors.

DETAILED DESCRIPTION:
This is a randomized, prospective, double-blind study. Randomization to Saxagliptin and placebo will be in a 2:1 fashion. Treatment duration will be approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   1. Before any study procedures are performed, subjects will have the details of the study described to them, and they will be given a written informed consent document to read. Then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel.
   2. Subjects must be able to communicate meaningfully with the investigator and legally competent to provide informed written consent.
2. Target Population

   1. Body mass index 27.5-37.5 kg/m2
   2. Stable body weight (not varying >10% during the last 6 months)
3. Age and Reproductive Status

   1. Men and women, ages 21 to 70 years.
   2. Women must be sterilized by hysterectomy or postmenopausal or on acceptable birth control if of childbearing potential.
   3. Women of childbearing potential (WOCBP) include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Post menopause is defined as:

      * Amenorrhea ≥12 consecutive months without another cause and a documented serum follicle stimulating hormone (FSH) level >35 mIU/mL, or
      * Women with irregular menstrual periods and a documented serum FSH level >35 mIU/mL, or NOTE: FSH level testing is not required for women ≥62 years old with amenorrhea of ≥1 year
      * Women on hormone replacement therapy (HRT) Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential.

Exclusion Criteria:

1. Sex and Reproductive Status

   1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period
   2. Women who are pregnant or breastfeeding
2. Target Disease Exceptions

   1. Gastrointestinal disease (including gastrectomy, chronic pancreatitis, bariatric surgery and gastroparesis)
   2. Hepatic disease (ALT, AST >2.5 times the upper limit of normal, high sensitivity CRP ≥1 mg/L)
   3. Kidney disease (serum creatinine >1.6 mg/dl, Creatinine Clearance 50 mL/min)
   4. Hypertension (blood pressure > 150/95 mmHg) at Screening for the mean of three consecutive readings performed in a sitting position after a 5-minute resting period. If treatment for hypertension has recently been initiated, subjects must be clinically stable for 4 weeks prior to Screening
   5. Cardiac disease (myocardial infarction within past year, clinically significant arrhythmia, unstable angina, congestive heart failure, or coronary artery bypass surgery within 1 year or expected to require coronary bypass surgery within 12 months of study entry).
3. Medical History and Concurrent Diseases

   1. Type 1 diabetes mellitus
   2. Type 2 diabetes mellitus
   3. History of diabetic ketoacidosis or hyperosmolar nonketotic coma
   4. Malignancy other than basal cell or squamous cell skin cancer
   5. Significant clinical allergic rhinitis or asthma, regularly requiring inhaled corticosteroids and/or antihistamines
4. Additional Laboratory Test Findings

   1. Hemoglobin <12 g/dl in men, <11 g/dl in women
   2. Abnormal prothrombin or partial thromboplastin time
   3. Clinically abnormal thyroid stimulating hormone (TSH)
   4. 2 hour glucose > 170mg/dl in standard oral glucose tolerance test (OGTT)
5. Allergies and Adverse Drug Reactions

   a. Subjects with a history of a serious hypersensitivity reaction to saxagliptin, such as anaphylaxis, angioedema,or exfoliative skin conditions.
6. Prohibited Treatments and/or Therapies

   1. Treatment with strong systemic cytochrome P450 3A4/5 (CYP 3A4/5) inhibitors
   2. Treatment with any of the following medications during screening or their expected use during the study: recent systemic glucocorticoids (for more than 2 weeks), any anti-hyperglycemic agents, antineoplastic agents, transplant medications, drugs for weight loss, niacin, fibrates, or anti-retroviral medications
   3. Treatment with beta-blockers, antihistamines or inhaled corticosteroids within 3 months prior to screening
   4. Start or change of hormonal replacement therapy within 3 months prior to screening
7. Other Exclusion Criteria

   1. Prisoners, or subjects who are involuntarily incarcerated
   2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness
   3. Currently abusing alcohol or drugs, or have a history of alcohol or drug abuse that in the investigator's opinion could cause the subject to be non-compliant; or have a general history of non-compliance with medications
   4. Any acute febrile illness within 2 weeks of screening with a temperature 100°F

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the secretion of cytokines/adipokines by adipose tissue | 6 weeks
  The primary objective is to determine whether 6 weeks of treatment with saxagliptin, compared to placebo, causes a reduction from baseline in the production and secretion of cytokines/adipokines by adipose tissue

SECONDARY OUTCOMES:
reduction from baseline in tissue measures of inflammation | 6 weeks
  The secondary objective is to determine whether 6 weeks of treatment with saxagliptin, compared to placebo, causes a reduction from baseline in reactive oxygen production, pro-inflammatory gene expression, toll-like receptor and nuclear factor-kappa B activation, and macrophage infiltration in adipose tissue of obese individuals
change in plasma postprandial lipids | 6 weeks
  We will also compare the change in postprandial lipids following a standard meal between placebo and saxagliptin
change in reactive hyperemic index | 6 weeks
  We will use peripheral artery tonometry to measure the change in endothelial function by measuring reactive hyperemic index

OTHER OUTCOMES:
change in percent arteriole dilation | 6 weeks
  Using arterioles isolated from tissue biopsies, we will measure dose related responses to distinct dilators

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Reaven, MD, Principal Investigator — Carl T. Hayden VA Medical Hospital
Locations (1):
- Carl T. Hayden VA Medical Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Subject to VA regulation.

REFERENCES:
- [Background] Kim SH, Liu A, Ariel D, Abbasi F, Lamendola C, Grove K, Tomasso V, Ochoa H, Reaven G. Effect of salsalate on insulin action, secretion, and clearance in nondiabetic, insulin-resistant individuals: a randomized, placebo-controlled study. Diabetes Care. 2014 Jul;37(7):1944-50. doi: 10.2337/dc13-2977. PMID 24963111